CLINICAL TRIAL: NCT03777202
Title: Efficacy of High Flow Nasal Oxygen During Sleep Endoscopy in Patients of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0923
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal oxygen during sleep endoscopy (Experimental): High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system during sleep endoscopy. Pulse oximetry will be monitored continuously. Otorhinolaryngologist will observe the degree of upper airway obstruction during sleep endoscopy.
  Interventions: Procedure: High-flow nasal oxygen
- Low-flow nasal oxygen during sleep endoscopy (Active Comparator): Low-flow nasal oxygen will be applied to the patients through nasal openings using conventional nasal cannula during sleep endoscopy. Pulse oximetry will be monitored continuously. Otorhinolaryngologist will observe the degree of upper airway obstruction during sleep endoscopy.
  Interventions: Procedure: Low-flow nasal oxygen

INTERVENTIONS:
Procedure: High-flow nasal oxygen — High-flow nasal oxygen will be applied to the patients using Optiflow system through nasal openings during sleep endoscopy. Pulse oximetry will be monitored continuously. Otorhinolaryngologist will observe the degree of upper airway obstruction during sleep endoscopy.
  Arms: High-flow nasal oxygen during sleep endoscopy
Procedure: Low-flow nasal oxygen — Low-flow nasal oxygen will be applied to the patients through nasal openings using conventional nasal cannula during sleep endoscopy. Pulse oximetry will be monitored continuously. Otorhinolaryngologist will observe the degree of upper airway obstruction during sleep endoscopy.
  Arms: Low-flow nasal oxygen during sleep endoscopy

SUMMARY:
The purpose of this study is to investigate the utility of high-flow nasal oxygen during sleep endoscopy in obstructive sleep apnea patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged over 19 years who are scheduled for sleep endoscopy

Exclusion Criteria:

* 1) basal skull fracture, 2) facial anomaly, 3) consciousness disorder, 4) Risk of aspiration, 5) necessity of awake fiberoptic intubation due to the large vocal cord mass, endotracheal tumor or bleeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
oxygen saturation value | For 15 minutes during sleep endoscopy. At Day 0.
  Pulse oximetry will be monitored continuously during sleep endoscopy. Oxygen saturation value will be recorded during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea